CLINICAL TRIAL: NCT06739967
Title: Speech and Language-Tailored Interventions for People With Primary Progressive Aphasia
Brief Title: Speech and Language Interventions for Italian People With PPA
Acronym: PPA-rehab
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 1767/CEL; PNRR-MCNT2-2023-12378220 (Other Grant/Funding Number: European Union-Next Generation EU-NRRP M6C2-Investment 2.1 Enhancement and strengthening of biomedical research in NHS)
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Primary Progressive Aphasia(PPA)
Keywords: Speech and language therapy; online intervention; Frontotemporal dementia; Alzheimer's disease; PPA; Communication Disorders; Neurodegenerative Diseases; Dementia
MeSH Terms: conditions — Aphasia, Primary Progressive; Communication Disorders; Frontotemporal Dementia; Neurodegenerative Diseases; Dementia | interventions — Behavior Therapy; Speech Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Speech and Language Tailored Interventions: Patients will receive three days a week for 5 weeks of 45 minute sessions of a tailored speech and language intervention
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — The SLT intervention will be entirely administered online through a web-based platform. While each of the treatments will engage semantics, phonology, and orthography, the protocols will be tailored relative to the characteristics of each PPA variant. Patients with svPPA and lvPPA will undergo a lexical retrieval training (LRT) intervention implemented using a training cascade.
  Patients with nfvPPA will undergo Video-implemented Script Training (VISTA), a choral reading approach training accurate production of functional scripts. The method is based on that implemented in American-English individuals with PPA and aims at improving grammar and motor aspects of speech production by taking advantage of repetitive practice and automaticity.
  Other Names: Speech and Language Therapy; SLT

SUMMARY:
Primary progressive aphasia (PPA) is an umbrella term used to refer to several clinical variants that manifest as an insidious deterioration of speech/language skills, usually due to frontotemporal lobar degeneration and/or Alzheimer's disease. Consensus criteria have been proposed by an international community regarding the sub-classification of PPA into three variants: (1) semantic variant PPA, characterized by impaired confrontation naming and single-word comprehension; (2) logopenic variant PPA), characterised by word-finding difficulties and sentence repetition deficits; and (3) non-fluent variant, characterised by agrammatism with or without apraxia of speech.

Speech and language therapists (SLTs) play a crucial role in the diagnostic process and in setting a therapeutic path along with monitoring the evolution of the clinical picture. Despite growing evidence supporting the benefits of speech-language intervention, the frequency with which individuals with PPA are referred for speech and language services, is suboptimal likely due to skepticism regarding the value of speech and language therapy in the context of neurodegeneration, the scarcity of SLTs with expertise in the treatment of PPA, the lack of awareness regarding the role of the SLT amongst referrers, and the geographical barriers that impede access to in-person speech and language services. In Italy, patients with PPA are rarely offered treatment options due to a lack of understanding of the disorder on the part of health professionals and erroneous assumptions regarding the utility of treatment in patients facing a worsening prognosis.

The primary aim of this pilot study is to develop tailored speech and language interventions for patients with different variants of PPA by addressing their linguistic and cognitive difficulties. Secondly, to explore the intervention's effect also on untreated tasks and assess the long-term maintenance of the proposed interventions by monitoring patients for up to six months. Finally, in each PPA variant, the investigators aim to investigate which variables among the sociodemographic, clinical, linguistic/cognitive, and brain MRI features at baseline predict successful clinical results, as well as which structural and functional brain changes are associated with speech and language improvements.

DETAILED DESCRIPTION:
A total of 30 PPA patients will be recruited, with a clinical and imaging-supported diagnosis of PPA according to the current diagnostic criteria, and MMSE>15. At the study entry (T0), all patients will undergo a clinical interview, a neurological and neuropsychological evaluation, and a speech and language assessment. All these visits will be repeated soon after the intervention (at week 5, W5), at 3 months (M3), and at 6 months (M6) post-intervention. Specifically, measures of patient's and caregivers' satisfaction and patients' functional communication abilities will be collected as primary outcomes. At baseline (T0) and after intervention (W5), all patients recruited at IRCCS San Raffaele and 40% of patients recruited at IRCCS Maugeri Clinical and Scientific Institute will also perform a brain structural and functional MRI. Thirty healthy controls, matched with PPA cases for age and sex, will be also recruited. Only at baseline (T0), all controls will undergo the same visits as the PPA patients, as well as the brain MRI scan. IRCCS Maugeri Clinical and Scientific Institute will be specifically in charge of the development of the SLT protocols, for the online administration of tailored speech and language interventions and for data analysis. IRCCS Ospedale San Raffaele Milano will be specifically in charge of brain structural and functional MRI acquisition, the definition of task-based functional MRI paradigms, and MRI analysis. This unit will also recruit and collect data on the entire sample of healthy controls. Brain structural and functional changes associated with SLT interventions using the most advanced MRI techniques will be investigated. The sociodemographic, clinical, language, speech, and MRI features obtained in patients will be processed through machine learning to develop a computation paradigm that better defines their prediction value for the intervention's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA according to the current clinical criteria (Gorno-Tempini et al., 2011)
* Mild PPA defined using the Progressive Aphasia Severity Scale (PASS)
* Age between 40 and 85 years
* Patients with Italian mother tongue
* Patients with the ability to sign the informed consent
* Patients with the ability to comply with the study procedures
* Patients with stable pharmacological treatment for at least 4 weeks.

Exclusion Criteria:

* Mini-Mental State Exam (MMSE) Score <15
* Presence of other neurological or psychiatric diseases, including cerebrovascular disease
* Severe and uncorrected hearing loss or visual disturbances
* Inability to repeat multi-syllable words (4 syllables)
* Concurrent participation in other pharmacological and non-pharmacological experimental studies

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary progressive aphasia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in measure of naming after Lexical Retrieval Training (LRT) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Number of correct spoken and written naming of trained and untrained items for patients undergoing the LRT treatment (lvPPA/svPPA)
Change in number of articulatory and grammatical errors | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  The percentage of script words produced correctly for VISTA for trained and untrained scripts.
Change in measures of patients and caregivers satisfaction and patients functional communication abilities | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  A Likert scale evaluating relevant categories of functional verbal communication skills in daily situations will be used. The score ranges from 0 - 30. High scores are more favorable, meaning that high scores indicate less interference in participation. The summary scores will be converted to IRT theta values (logit scale). On the logit scale, scores range from -3.0 to +3.0 with 0 logits representing the mean for the calibration sample. High scores are preferable.
Change on untrained probes within each clinical variant | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Number of untrained items correctly identified

SECONDARY OUTCOMES:
Change in measure of oral production as assessed by Picture description subtests | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  To examine the informativeness and efficiency of communication from the connected speech sampled with the Nicholas and Brookshire (1993) picture description task and the Screening for Aphasia in Neurodegeneration (SAND) picture task.
Change in measure of quality of life as assessed by Communication Outcome After Stroke (COAST) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Communication Outcome After Stroke (COAST) is a measure of the functional communication in daily activities and of the impact of the quality of life point of view of aphasia patient (COAST total score range: min= 0, max= 80, higher score=better outcome) and their carer (Carer COAST total score range: min= 0, max= 80, higher score=better outcome)
Change in measure of naming as assessed by Picture Naming subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Picture Naming subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 14, higher score=better outcome), living score (score range: min= 0, max= 7, higher score=better outcome) and non-living score (score range: min= 0, max= 7, higher score=better outcome).
Change in measure of comprehension as assessed by Auditory sentence comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Auditory sentence comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND): total score range: min= 0, max= 8, higher score=better outcome.
Change in measure of comprehension as assessed by Single-word comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Single-word comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 12, higher score=better outcome), living score (score range: min= 0, max= 6, higher score=better outcome) and non-living score (score range: min= 0, max= 6, higher score=better outcome).
Change in measure of repetition as assessed by Repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 10, higher score=better outcome), words score (score range: min= 0, max= 6, higher score=better outcome) and non-words score (score range: min= 0, max= 4, higher score=better outcome).
Change in measure of repetition as assessed by Sentence repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Sentence repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 6, higher score=better outcome), predictable sentences score (score range: min= 0, max= 3, higher score=better outcome) and unpredictable sentences score (score range: min= 0, max= 3, higher score=better outcome).
Change in measure of reading as assessed by Reading subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Reading subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 16, higher score=better outcome), words score (score range: min= 0, max= 12, higher score=better outcome) and non-words score (score range: min= 0, max= 4, higher score=better outcome).
Change in measure of writing as assessed by Writing subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Writing subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides Information Units score (score range: min= 0, max= 6, higher score=better outcome), total number of words score (score range: min= 0, max= no limits, higher score=better outcome), number of nouns/total number of words score (score range: min= 0, max= 1, higher score=better outcome), number of verbs/total number of words (score range: min= 0, max= 1, higher score=better outcome), number of correct syntactic structures/total number of syntactic structures score (score range: min= 0, max= 1, higher score=better outcome), number of orthographic errors score (score range: min= 0, max= no limits, higher score=worse outcome), number of lexico-semantic errors/number of words score (score range: min= 0, max= 1, higher score=worse outcome).
Change in measure of semantics as assessed by Semantic association subtest from Screening for Aphasia in NeuroDegeneration (SAND) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Semantic association subtest from Screening for Aphasia in NeuroDegeneration (SAND): total score range: min= 0, max= 4, higher score=better outcome.
Change in measure of naming as assessed by Subtest from CAGI battery | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Naming subtest from CAGI: score range: min= 0, max= 48, higher score=better outcome.
Change in measure of comprehension as assessed by Single-word comprehension subtest from CAGI | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Single-word comprehension subtest from CAGI: score range: min= 0, max= 48, higher score=better outcome.
Change in measure of Sentence Production as measured by Northwestern Anagram Test-Italian (Nat-I) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  The NAT-I is a 22-item test: score range: min= 0, max= 22, higher score=better outcome.
Change in measure of comprehension as assessed by Sentence Comprehension Task | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Sentence Comprehension Task: total score range: min= 0, max= 48, higher score=better outcome.
Change in in measure of verb and sentence processing as measured by the Italian version of the Northwestern Assessment of Verbs and Sentences (NAVS-I) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  NAVS-I encompasses three subtests: Verb Naming Task (VNT), Verb Comprehension Task (VCT), and Argument Structure Production Task (ASPT).
Change in measure of semantics as assessed by Semantic association Test (SAT) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  SAT: total score range: min= 0, max= 76, higher score=better outcome.
Change in measure of repetition as assessed by Repetition subtest from Esame Neuropsicologico per l'Afasia (ENPA) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Repetition subtest from ENPA: score range: min= 0, max= 15, higher score=better outcome.
Change in measure of repetition as assessed by Repetition subtest from Aachener Aphasie Test (AAT) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Repetition subtest from AAT: score range: min= 0, max= 150, higher score=better outcome.
Changes in measures of motor speech as assessed by the Motor Speech Evaluation (MSE) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Motor Speech Evaluation (MSE) score range: min= 0, max= 30, higher score=better outcome.
Change in measures of Verbal fluency as measured by Phonemic Fluency Test and Semantic Fluency Test | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Phonemic Fluency Test: higher score= better outcome. Semantic Fluency Test: higher score= better outcome.
Change in measure of global cognitive impairment as assessed by Mini Mental State Examination (MMSE) | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Mini Mental State Examination (MMSE): score range: min= 0, max= 30, higher score=better outcome.
Change in dementia severity as assessed by Frontotemporal Dementia- Clinical Dementia Rating Scale (FTD-CDR)- Sum of Boxes | From enrollment to the end of treatment at 5 weeks, 3 Months and 6 Months
  Frontotemporal Dementia- Clinical Dementia Rating Scale (FTD-CDR)- Sum of Boxes (score range: min= 0, max= 24, higher score=worse outcome).
Structural MRI scan | At baseline, from enrollment to the end of treatment at 5 weeks
  Measure of global and regional volumes of interest (such as whole brain and temporal lobes). Tissue health (from structural scan) will be obtained at baseline to investigate neural predictors of treatment outcome.
Functional MRI scan | At baseline, from enrollment to the end of treatment at 5 weeks
  Task-based activation location (from functional MRI scans) will be obtained at baseline to investigate neural predictors of treatment outcome. Connectivity between brain regions measured using diffusion tensor MRI and resting state functional MRI.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituti Clinici Scientifici Maugeri IRCCS, Bari
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No
Privacy Concerns: Protecting the confidentiality of participants is a priority. Sharing IPD could risk the exposure of sensitive personal information.

REFERENCES:
- [Background] Tippett DC, Hillis AE, Tsapkini K. Treatment of Primary Progressive Aphasia. Curr Treat Options Neurol. 2015 Aug;17(8):362. doi: 10.1007/s11940-015-0362-5. PMID 26062526
- [Background] Grossman M. Primary progressive aphasia: clinicopathological correlations. Nat Rev Neurol. 2010 Feb;6(2):88-97. doi: 10.1038/nrneurol.2009.216. PMID 20139998
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Mesulam MM. Primary progressive aphasia--differentiation from Alzheimer's disease. Ann Neurol. 1987 Oct;22(4):533-4. doi: 10.1002/ana.410220414. No abstract available. PMID 3324947
- [Background] Volkmer A, Rogalski E, Henry M, Taylor-Rubin C, Ruggero L, Khayum R, Kindell J, Gorno-Tempini ML, Warren JD, Rohrer JD. Speech and language therapy approaches to managing primary progressive aphasia. Pract Neurol. 2020 Apr;20(2):154-161. doi: 10.1136/practneurol-2018-001921. Epub 2019 Jul 29. PMID 31358572
- [Background] Battista P, Piccininni M, Montembeault M, Messina A, Minafra B, Miller BL, Henry ML, Gorno Tempini ML, Grasso SM. Access, referral, service provision and management of individuals with primary progressive aphasia: A survey of speech-language therapists in Italy. Int J Lang Commun Disord. 2023 Jul-Aug;58(4):1046-1060. doi: 10.1111/1460-6984.12843. Epub 2023 Jan 13. PMID 36636857
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651